CLINICAL TRIAL: NCT05551507
Title: A Phase Ib/II, Open-label Clinical Study to Evaluate the Safety, Tolerability and Antitumor Activities of IN10018 in Combination With Standard Chemotherapy in Subjects With High-grade Serous Epithelial Ovarian Cancer
Brief Title: IN10018 in Combination With Standard Chemotherapy in High-grade Serous Epithelial Ovarian Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN10018-006
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Platinum-resistant Ovarian Cancer
MeSH Terms: interventions — 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IN10018 in combination with PLD (Experimental): IN10018 in combination with PLD in platinum-resistant recurrent epithelial ovarian cancer, fallopian tube cancer or primary peritoneum cancer with the subtype limited to high-grade serous carcinoma subjects.
  Interventions: Drug: IN10018 in combination with PLD

INTERVENTIONS:
Drug: IN10018 in combination with PLD — IN10018 in combination with PLD to treat subjects with platinum-resistant recurrent ovarian cancer
  Other Names: IN10018 add on to PLD treatment

SUMMARY:
This is a phase Ib/II, open label clinical study to evaluate the safety, tolerability and antitumor activities of IN10018 in combination with standard chemotherapy in subjects with high-grade serous ovarian cancer (including fallopian tube cancer and primary peritoneum cancer, collectively defined as ovarian cancer).

DETAILED DESCRIPTION:
Study will evaluate IN10018 in combination with pegylated liposomal doxorubicin (PLD) in subjects with platinum-resistant recurrent ovarian cancer. All the subjects will receive combination therapy until documented progressive disease or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign informed consent(s). Signed informed consent must be obtained before any study specific procedures, except those procedures used as institutional standard of care falling into the protocol specified window and fulfilling study specific requirements such as tumor imaging.
2. Female subjects ≥ 18 years at the time of signing informed consent.
3. Histologically confirmed epithelia ovarian cancer, fallopian tube cancer or primary peritoneum cancer with the subtype limited to high-grade serous carcinoma (HGSC) only.
4. Subjects with platinum-resistant disease, defined as having relapsed or progressed between 1- 6 months after completion of prior platinum-based therapy (at least 4 cycles).
5. Have maximum total of 5 prior lines of systemic therapy and maximum 2 prior lines of systemic therapy following diagnosis of platinum-resistance.
6. At least one measurable lesion can be accurately measured per RECIST 1.1 as assessed by investigator.
7. ECOG performance status of 0 or 1.
8. Life expectancy of at least 3 months as assessed by investigator.
9. Availability of archival or fresh (newly obtained) tumor tissue sample during Screening Phase: Fresh tumor tissue sample obtained after most recent relapse or progression is preferred; if no sample or not sufficient number of slides can be provided or collected, a joint decision between Sponsor and investigator is needed for the enrollment of this subject.
10. Must have recovered from all AEs due to previous therapies to ≤ Grade 1 (CTCAE 5.0) or stable status as assessed by investigator.
11. Adequate bone marrow, liver, renal, and coagulation function within 5 days prior to first dose of study treatment.
12. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP) . OR
    * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and through 3 months after the last dose of study treatment.

Exclusion Criteria:

1. Has had major surgery or significant traumatic injury within 28 days prior to first dose of study treatment, or diagnostic biopsies within 14 days prior to first dose of study treatment.
2. Has received prior systemic anticancer therapy including investigational agents, such as within 14 days or less than 5 half-lives (whichever is shorter) of chemotherapy or targeted therapy, or within 28 days of immunotherapy, prior to first dose of study treatment.
3. Has received prior radiotherapy within 14 days prior to first dose of study treatment.
4. Has received prior treatment of any FAK inhibitor or prior treatment of PLD.
5. Has a known previous or concurrent cancer that is distinct in primary site or histology from current ovarian cancer within 3 years prior to first dose of study treatment, except for curatively treated cancers such as cervical carcinoma in situ.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
7. Has a history of major cardiovascular, cerebrovascular or thromboembolic diseases (e.g., congestive heart failure, acute myocardial infarction, unstable angina, stroke, transient ischemic attack, deep vein thrombosis or pulmonary embolism) within 6 months before first dose of study treatment, or has any of the following abnormality:

   * QTc interval > 480 msec;
   * Left ventricular ejection fraction (LVEF) < 50%;
   * New York Heart Association (NYHA) functional classification ≥ Grade 2；
   * Clinically significant arrhythmia;
   * Uncontrolled hypertension;
   * Other clinically significant heart diseases.
8. Has known uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage. Note: A small amount of ascites that can only be detected by imaging examination is allowed.
9. Has malabsorption syndrome or inability to take oral drugs.
10. Has clinically significant gastrointestinal abnormalities including uncontrolled gastrointestinal inflammatory lesions (Crohn's disease, or ulcerative colitis in active) or uncontrolled gastrointestinal bleeding.
11. Has an active infection requiring systemic therapy within 14 days prior to the first dose of study treatment.
12. Has known human immunodeficiency virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority and/or site.
13. Has known active Hepatitis B or Hepatitis C virus infection. Note: No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority and/or site.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.
16. Known allergy or hypersensitivity to IN10018 or PLD, or their ingredients.
17. Has received prior cumulative anthracycline dose of 550 mg/m2 or more.
18. Has received systemic treatment of CYP3A4, CYP2D6 or P-gp strong inhibitors/inducers within 14 days prior to the first dose of study treatment, or anticipation of the systemic treatment of these drugs during Treatment Phase.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events per NCI-CTCAE version 5.0. | Up to 24 months
  Incidence of Treatment-Emergent Adverse Events per NCI-CTCAE version 5.0.
Recommended phase 2 dose (RP2D) of the combination. | Up to 2 months
  Defined based on the incidence of dose limiting toxicities (DLTs).
Objective response rate (ORR) as assessed by investigator. | Up to 24 months
  ORR is defined as the proportion of subjects with complete response (CR) and partial response (PR), as assessed by investigator per RECIST 1.1.

SECONDARY OUTCOMES:
Objective response rate (ORR) as assessed by blinded independent central review (BICR). | Up to 24 months
  ORR is defined as the proportion of subjects with complete response (CR) and partial response (PR), as assessed by BICR per RECIST 1.1.
Duration of response (DOR) as assessed by investigator and BICR. | Up to 24 months
  DOR is defined as the time from the first occurrence of objective response to disease progression or death from any cause (whichever occurs first), as assessed by investigator and BICR per RECIST 1.1.
Disease control rate (DCR) as assessed by investigator and BICR. | Up to 24 months
  DCR is defined as the proportion of subjects with CR or PR, or stable disease, as assessed by investigator and BICR per RECIST 1.1.
Progression free survival (PFS) as assessed by investigator and BICR. | Up to 24 months
  PFS is defined as the time from start of treatment to the first occurrence of disease progression or death from any cause (whichever occurs first), as assessed by investigator and BICR per RECIST 1.1.
Overall survival (OS) | Up to 24 months
  OS is defined as the time from start of treatment to death from any cause.
CA 125 response rate per Gynecological Cancer Inter-group (GCIG) criteria. | Up to 24 months
  CA 125 response rate per GCIG criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (7):
- China (7):
  - Anyang Cancer Hospital, Anyang
  - Cancer Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing
  - Hunan Cancer Hospital, Changsha
  - Fujian Cancer Hospital, Fuzhou
  - Affiliated Obstetrics and Gynecology Hospital of Zhejiang University, Hangzhou
  - Tianjin Cancer Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No